CLINICAL TRIAL: NCT01786512
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter, Dose Escalation Study to Select and Evaluate an Oral Modified Release Formulation of Omecamtiv Mecarbil in Subjects With Heart Failure and Left Ventricular Systolic Dysfunction
Brief Title: COSMIC-HF - Chronic Oral Study of Myosin Activation to Increase Contractility in Heart Failure
Acronym: COSMIC-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110151; 2012-000327-40 (EudraCT Number)
Record Dates: First submitted 2013-01-18; First posted 2013-02-08 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Modified Release Oral Formulation; Left Ventricular Systolic Dysfunction; Chronic Heart Failure; History of Chronic Heart Failure; Left Ventricular Ejection Fraction; Pharmacokinetics; Echocardiogram
Keywords: Pharmacokinetics; Omecamtiv mecarbil; AMG 423; Double-blind; Randomized; Placebo-controlled; Oral forumlation; CK-1827452; Cardiac myosin activator
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Dose-escalation Cohort 1: Placebo (Placebo Comparator): Participants received placebo tablets twice a day (BID) for 7 days.
  Interventions: Drug: Placebo
- Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 (Experimental): Participants received 25 mg omecamtiv mecarbil (OM) Matrix F1 (M-F1) tablets twice a day for 7 days.
  Interventions: Drug: Omecamtiv Mecarbil Matrix F1 Formulation
- Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 (Experimental): Participants received 25 mg omecamtiv mecarbil Matrix F2 (M-F2) tablets twice a day for 7 days.
  Interventions: Drug: Omecamtiv Mecarbil Matrix F2 Formulation
- Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 (Experimental): Participants received 25 mg omecamtiv mecarbil swellable core technology F2 (SCT-F2) tablets twice a day for 7 days.
  Interventions: Drug: Omecamtiv Mecarbil Swellable Core Technology F2
- Dose-escalation Cohort 2: Placebo (Placebo Comparator): Participants received placebo tablets twice a day for 7 days.
  Interventions: Drug: Placebo
- Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 (Experimental): Participants received 50 mg omecamtiv mecarbil M-F1 tablets twice a day for 7 days.
  Interventions: Drug: Omecamtiv Mecarbil Matrix F1 Formulation
- Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 (Experimental): Participants received 50 mg omecamtiv mecarbil M-F2 tablets twice a day for 7 days.
  Interventions: Drug: Omecamtiv Mecarbil Matrix F2 Formulation
- Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2 (Experimental): Participants received 50 mg omecamtiv mecarbil SCT-F2 tablets twice a day for 7 days.
  Interventions: Drug: Omecamtiv Mecarbil Swellable Core Technology F2
- Expansion Phase: Placebo (Placebo Comparator): Participants received placebo tablets twice a day for 20 weeks.
  Interventions: Drug: Placebo
- Expansion Phase: Omecamtiv Mecarbil 25 mg M-F1 (Experimental): Participants received 25 mg omecamtiv mecarbil M-F1 tablets twice a day for 20 weeks.
  Interventions: Drug: Omecamtiv Mecarbil Matrix F1 Formulation
- Expansion Phase: OM M-F1 PK-based Titration (Experimental): All participants received 25 mg omecamtiv mecarbil M-F1 tablets twice a day. At week 8 the dose escalated to 50 mg twice a day if the week 2 predose plasma concentration of OM was less than the predefined cutoff of 200 ng/mL.
  Interventions: Drug: Omecamtiv Mecarbil Matrix F1 Formulation

INTERVENTIONS:
Drug: Omecamtiv Mecarbil Matrix F1 Formulation — Modified release tablets for oral administration
  Other Names: AMG 423; CK-1827452
  Arms: Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1; Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1; Expansion Phase: OM M-F1 PK-based Titration; Expansion Phase: Omecamtiv Mecarbil 25 mg M-F1
Drug: Omecamtiv Mecarbil Matrix F2 Formulation — Modified release tablets for oral administration
  Other Names: AMG 423; CK-1827452
  Arms: Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2; Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2
Drug: Placebo — Modified release tablets matching to omecamtiv mecarbil
  Arms: Dose-escalation Cohort 1: Placebo; Dose-escalation Cohort 2: Placebo; Expansion Phase: Placebo
Drug: Omecamtiv Mecarbil Swellable Core Technology F2 — Modified release tablets for oral administration
  Other Names: AMG 423; CK-1827452
  Arms: Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2; Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2

SUMMARY:
The primary objectives of this study are (i) to select an oral modified release (MR) formulation and dose of omecamtiv mecarbil for chronic twice daily (BID) dosing in adults with heart failure and left ventricular systolic dysfunction and (ii) to characterize its pharmacokinetics (PK) over 20 weeks of treatment.

DETAILED DESCRIPTION:
Omecamtiv mecarbil (AMG 423, CK-1827452) is a novel small molecule that increases cardiac contractility by selectively and directly activating the enzymatic domain of cardiac myosin heavy chain, the force-generating motor protein of the cardiac sarcomere. This is a randomized, placebo-controlled, multicenter, phase 2 study, consisting of a dose escalation phase to select 1 of 3 omecamtiv mecarbil oral formulations in 2 dose escalation cohorts, followed by an expansion phase to evaluate 20 weeks of administration of the selected omecamtiv mecarbil formulation at 2 target dose levels, compared with placebo.

This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic heart failure (HF), defined as requiring treatment for HF for a minimum of 4 weeks prior to screening
* Treated with stable, optimal pharmacological therapy for ≥ 4 weeks
* History of left ventricular ejection fraction (LVEF) ≤ 40%
* Elevated N-terminal prohormone B-type natriuretic peptide (NT-proBNP)

Exclusion criteria:

* Severe uncorrected valvular heart disease
* Hospitalization within 30 days prior to enrollment
* Hypertrophic obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, or clinically significant congenital heart disease
* Acute myocardial infarction, unstable angina or persistent angina at rest within 30 days prior to randomization
* Systolic blood pressure > 160 mmHg or < 90 mmHg or diastolic blood pressure > 90 mmHg
* Total bilirubin ≥ 2 x upper limit of normal (ULN); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 x ULN
* Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m^2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2013-02-26 (Actual); Primary Completion 2015-07-22 (Actual); Study Completion 2015-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (95):
- United States (37):
  - Research Site, Mobile, Alabama
  - Research Site, Costa Mesa, California
  - Research Site, Fresno, California
  - Research Site, Inglewood, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Thousand Oaks, California
  - Research Site, Tustin, California
  - Research Site, Danbury, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Atlantis, Florida
  - Research Site, Aventura, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Auburn, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cortlandt Manor, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Australia (2):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Nedlands, Western Australia
- Belgium (5):
  - Research Site, Antwerp
  - Research Site, Bonheiden
  - Research Site, Ghent
  - Research Site, Ieper
  - Research Site, Liège
- Bulgaria (7):
  - Research Site, Kazanlak
  - Research Site, Pazardzhik
  - Research Site, Plovdiv
  - Research Site, Sandanski
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
- Canada (9):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Svitavy
  - Research Site, Teplice
- Germany (5):
  - Research Site, Bad Krozingen
  - Research Site, Bad Nauheim
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Greifswald
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Jászberény
  - Research Site, Zalaegerszeg
- Italy (3):
  - Research Site, Brescia
  - Research Site, Pavia
  - Research Site, Verona
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Netherlands (3):
  - Research Site, Amersfoort
  - Research Site, Groningen
  - Research Site, Utrecht
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Kłodzko
  - Research Site, Lublin
  - Research Site, Ruda Śląska
  - Research Site, Warsaw
  - Research Site, Wroclaw
- United Kingdom (7):
  - Research Site, Dudley
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London

REFERENCES:
- [Background] Teerlink JR, Felker GM, McMurray JJ, Solomon SD, Adams KF Jr, Cleland JG, Ezekowitz JA, Goudev A, Macdonald P, Metra M, Mitrovic V, Ponikowski P, Serpytis P, Spinar J, Tomcsanyi J, Vandekerckhove HJ, Voors AA, Monsalvo ML, Johnston J, Malik FI, Honarpour N; COSMIC-HF Investigators. Chronic Oral Study of Myosin Activation to Increase Contractility in Heart Failure (COSMIC-HF): a phase 2, pharmacokinetic, randomised, placebo-controlled trial. Lancet. 2016 Dec 10;388(10062):2895-2903. doi: 10.1016/S0140-6736(16)32049-9. Epub 2016 Dec 1. PMID 27914656
- [Derived] Biering-Sorensen T, Minamisawa M, Liu J, Claggett B, Papolos AI, Felker GM, McMurray JJV, Legg JC, Malik FI, Honarpour N, Kurtz CE, Teerlink JR, Solomon SD. The effect of the cardiac myosin activator, omecamtiv mecarbil, on right ventricular structure and function in chronic systolic heart failure (COSMIC-HF). Eur J Heart Fail. 2021 Jun;23(6):1052-1056. doi: 10.1002/ejhf.2181. Epub 2021 May 5. No abstract available. PMID 33826209
- [Derived] Biering-Sorensen T, Minamisawa M, Claggett B, Liu J, Felker GM, McMurray JJV, Malik FI, Abbasi S, Kurtz CE, Teerlink JR, Solomon SD. Cardiac Myosin Activator Omecamtiv Mecarbil Improves Left Ventricular Myocardial Deformation in Chronic Heart Failure: The COSMIC-HF Trial. Circ Heart Fail. 2020 Dec;13(12):e008007. doi: 10.1161/CIRCHEARTFAILURE.120.008007. Epub 2020 Nov 12. No abstract available. PMID 33176443
- [Derived] Felker GM, Solomon SD, McMurray JJV, Cleland JGF, Abbasi SA, Malik FI, Zhang H, Globe G, Teerlink JR; COSMIC-HF Investigators. Effects of Omecamtiv Mecarbil on Symptoms and Health-Related Quality of Life in Patients With Chronic Heart Failure: Results From the COSMIC-HF Study. Circ Heart Fail. 2020 Dec;13(12):e007814. doi: 10.1161/CIRCHEARTFAILURE.120.007814. Epub 2020 Nov 12. PMID 33176437
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic heart failure treated with stable, optimal pharmacological therapy for ≥ 4 weeks were enrolled from February 2013 to March 2015 at 86 centers in 13 countries in Europe, Australia, and North America.
  The study consisted of a dose-escalation phase to select 1 of 3 omecamtiv mecarbil (OM) oral formulations in 2 dose cohorts, and an expansion phase to evaluate 20 weeks of treatment with the selected formulation at 2 target dose levels, compared with placebo.
Pre-assignment Details: In each of the dose-escalation cohorts participants were randomized equally to receive 1 of the 3 formulations of OM or placebo. In the expansion phase participants were randomized equally to receive 25 mg oral OM twice daily (fixed-dose group), 25 mg oral OM twice daily titrated up to 50 mg twice daily (pharmacokinetic-titration group), or oral placebo. Randomization in both phases was stratified by presence or absence of atrial fibrillation/flutter.
Groups:
- Expansion Phase: Omecamtiv Mecarbil 25 mg: Participants received 25 mg omecamtiv mecarbil M-F1 tablets twice a day for 20 weeks.
- Expansion Phase: OM PK-based Titration: Participants received 25 mg omecamtiv mecarbil M-F1 tablets twice a day. At week 8 the dose escalated to 50 mg twice a day if the week 2 predose plasma concentration of OM was less than the predefined cutoff of 200 ng/mL.
Period: Overall Study
Arm/Group | Dose-escalation Cohort 1: Placebo | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Placebo | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2 | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Started | 11 | 11 | 14 | 13 | 10 | 11 | 12 | 14 | 149 | 150 | 149
Received Study Treatment | 11 | 10 | 14 | 13 | 10 | 11 | 11 | 14 | 149 | 150 | 146
Completed | 11 | 10 | 14 | 13 | 10 | 11 | 11 | 14 | 145 | 145 | 137
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 5 | 12
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Decision by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-escalation Cohort 1: Placebo | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Placebo | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2 | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration | Total
Number analyzed (Participants) | 11 | 11 | 14 | 13 | 10 | 11 | 12 | 14 | 149 | 150 | 149 | 544
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (4.6) | 67.7 (11.4) | 65.3 (8.8) | 66.7 (8.7) | 62.1 (9.3) | 65.1 (7.0) | 63.8 (11.6) | 64.3 (11.5) | 63.7 (9.7) | 62.8 (10.2) | 62.7 (11.7) | 63.4 (10.4)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 3 | 4 | 7 | 5 | 5 | 6 | 5 | 6 | 82 | 81 | 76 | 280
  65 - 74 years | 8 | 4 | 4 | 6 | 5 | 4 | 4 | 5 | 46 | 52 | 50 | 188
  75 - 84 years | 0 | 3 | 3 | 2 | 0 | 1 | 3 | 3 | 21 | 17 | 23 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 1 | 3 | 3 | 4 | 2 | 30 | 23 | 24 | 97
  Male | 9 | 9 | 11 | 12 | 7 | 8 | 8 | 12 | 119 | 127 | 125 | 447
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 7 | 4 | 17
  Not Hispanic or Latino | 11 | 10 | 14 | 12 | 9 | 11 | 11 | 14 | 147 | 143 | 145 | 527
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Black or African American | 3 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 11 | 5 | 8 | 34
  Mixed Race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 7 | 10 | 14 | 12 | 10 | 8 | 11 | 12 | 136 | 142 | 140 | 502
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Stratification Factor - Atrial Fibrillation/Flutter at Randomization [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 3 | 2 | 0 | 1 | 2 | 3 | 32 | 32 | 32 | 107
  No | 11 | 11 | 11 | 11 | 10 | 10 | 10 | 11 | 117 | 118 | 117 | 437

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase: Maximum Observed Plasma Concentration (Cmax) of Omecamtiv Mecarbil Following the Last Dose (Day 7)
Time Frame: Day 7 at predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours, and 7 days post-dose.
Population: The pharmacokinetic analysis set (PKAS) included all randomized participants who received at least 1 dose of OM and had at least 1 evaluable OM PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2
Number analyzed (Participants) | 10 | 14 | 13 | 10 | 11 | 14
ng/mL | 193 (58.8) | 201 (94.4) | 171 (53.8) | 492 (115) | 502 (138) | 601 (204)

2. Primary Outcome: Dose Escalation Phase: Time to Maximum Observed Plasma Concentration (Tmax) of Omecamtiv Mecarbil Following the Last Dose (Day 7)
Time Frame: Day 7 at predose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours, and 7 days post-dose.
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2
Number analyzed (Participants) | 10 | 14 | 13 | 10 | 11 | 14
hours | 3.9 (4.4) | 2.0 (1.2) | 4.2 (1.9) | 2.6 (2.4) | 2.2 (1.8) | 4.6 (2.3)

3. Primary Outcome: Dose Escalation Phase: Plasma Concentration of Omecamtiv Mecarbil Prior to Dosing on Day 7
Time Frame: Day 7 at predose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2
Number analyzed (Participants) | 10 | 14 | 13 | 10 | 11 | 14
ng/mL | 157 (63.7) | 137 (56.8) | 134 (54.7) | 376 (170) | 395 (108) | 476 (234)

4. Primary Outcome: Dose Escalation Phase: Area Under the Plasma Concentration-time Curve for a Dosing Interval of 12 Hours Post Dose (AUC12) for Omecamtiv Mecarbil
Time Frame: Day 7 at predose and at 0.5, 1, 2, 3, 4, 6, 8, and 12 hours post-dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2
Number analyzed (Participants) | 10 | 14 | 13 | 10 | 11 | 14
ng*hr/mL | 2030 (658) | 2000 (1020) | 1740 (586) | 5070 (1060) | 5010 (1160) | 6550 (2340)

5. Primary Outcome: Expansion Phase: Plasma Concentration of Omecamtiv Mecarbil Prior to Dosing
Time Frame: Predose (before morning dose) at weeks 2, 8, 12, 16, and 20
Population: Pharmacokinetic analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 147 | 141
ng/mL
  Week 2: number analyzed (Participants) | 142 | 136
  Week 2 | 174 (62.2) | 179 (68.8)
  Week 8: number analyzed (Participants) | 134 | 130
  Week 8 | 156 (69.1) | 161 (74.4)
  Week 12: number analyzed (Participants) | 135 | 126
  Week 12 | 165 (67.9) | 263 (116)
  Week 16: number analyzed (Participants) | 124 | 119
  Week 16 | 155 (69.0) | 240 (120)
  Week 20: number analyzed (Participants) | 131 | 121
  Week 20 | 149 (71.2) | 239 (118)

6. Primary Outcome: Expansion Phase: Maximum Observed Plasma Concentration of Omecamtiv Mecarbil
Time Frame: Weeks 2 and 12 at predose and 1, 2, 4, 6, and 8 hours post-dose.
Population: Pharmacokinetic analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 147 | 141
ng/mL
  Week 2: number analyzed (Participants) | 146 | 141
  Week 2 | 212 (70.4) | 212 (81.0)
  Week 12: number analyzed (Participants) | 137 | 127
  Week 12 | 200 (71.1) | 318 (129)

7. Secondary Outcome: Expansion Phase: Change From Baseline in Systolic Ejection Time (SET) at Week 20
Description: Systolic ejection time was measured using echocardiography. Least squares means are from a repeated measures model including treatment group, stratification factor, scheduled visit, interaction of treatment with scheduled visit and the baseline value as covariates.
Time Frame: Baseline and week 20
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug. The repeated-measures model included all observed values.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 149 | 150 | 146
seconds | 0.0000 (0.0025) | 0.0112 (0.0024) | 0.0250 (0.0026)
Statistical Analysis 1: Comparison: Expansion Phase: Placebo vs Expansion Phase: Omecamtiv Mecarbil 25 mg; Test type: Other; p = 0.0007, Repeated Measures; Treatment difference = 0.0112, 95% CI 2-sided [0.0047 to 0.0176], Standard Error of Mean 0.0033 — Repeated measures model includes treatment group, stratification factor, scheduled visit, interaction of treatment with scheduled visit and the baseline value as covariates
Statistical Analysis 2: Comparison: Expansion Phase: Placebo vs Expansion Phase: OM PK-based Titration; Test type: Other; p < 0.0001, Repeated Measures; Treatment difference = 0.0250, 95% CI 2-sided [0.0184 to 0.0315], Standard Error of Mean 0.0033 — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Expansion Phase: Change From Baseline in Stroke Volume at Week 20
Description: Stroke volume was measured using echocardiography. Least squares means are from a repeated measures model including treatment group, stratification factor, scheduled visit, interaction of treatment with scheduled visit and the baseline value as covariates.
Time Frame: Baseline and week 20
Population: The full analysis set included all randomized participants who received at least 1 dose of study drug. The repeated-measures model included all observed values.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 149 | 150 | 146
mL | -1.05 (1.18) | 3.53 (1.16) | 2.58 (1.19)
Statistical Analysis 1: Comparison: Expansion Phase: Placebo vs Expansion Phase: Omecamtiv Mecarbil 25 mg; Test type: Other; p = 0.0036, Repeated Measures; Treatment difference = 4.58, 95% CI 2-sided [1.50 to 7.65], Standard Error of Mean 1.56 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Expansion Phase: Placebo vs Expansion Phase: OM PK-based Titration; Test type: Other; p = 0.0217, Repeated Measures; Treatment difference = 3.63, 95% CI 2-sided [0.53 to 6.72], Standard Error of Mean 1.57 — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Expansion Phase: Change From Baseline in Left Ventricular End Systolic Diameter (LVESD) at Week 20
Description: LVESD was measured using echocardiography. Least squares means are from a repeated measures model including treatment group, stratification factor, scheduled visit, interaction of treatment with scheduled visit and the baseline value as covariates.
Time Frame: Baseline and week 20
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 149 | 150 | 146
cm | -0.242 (0.043) | -0.322 (0.044) | -0.421 (0.045)
Statistical Analysis 1: Comparison: Expansion Phase: Placebo vs Expansion Phase: Omecamtiv Mecarbil 25 mg; Test type: Other; p = 0.1732, Repeated Measures; Treatment difference = -0.079, 95% CI 2-sided [-0.194 to 0.035], Standard Error of Mean 0.058 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Expansion Phase: Placebo vs Expansion Phase: OM PK-based Titration; Test type: Other; p = 0.0027, Repeated Measures; Treatment difference = -0.179, 95% CI 2-sided [-0.295 to -0.062], Standard Error of Mean 0.059 — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Expansion Phase: Change From Baseline in Left Ventricular End Diastolic Diameter (LVEDD) at Week 20
Description: LVEDD was measured using echocardiography. Least squares means are from a repeated measures model including treatment group, stratification factor, scheduled visit, interaction of treatment with scheduled visit and the baseline value as covariates.
Time Frame: Baseline and week 20
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 149 | 150 | 146
cm | 0.089 (0.038) | 0.023 (0.038) | -0.040 (0.040)
Statistical Analysis 1: Comparison: Expansion Phase: Placebo vs Expansion Phase: Omecamtiv Mecarbil 25 mg; Test type: Other; p = 0.1899, Repeated Measures; Treatment difference = -0.067, 95% CI 2-sided [-0.166 to 0.033], Standard Error of Mean 0.051 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Expansion Phase: Placebo vs Expansion Phase: OM PK-based Titration; Test type: Other; p = 0.0128, Repeated Measures; Treatment difference = -0.129, 95% CI 2-sided [-0.231 to -0.028], Standard Error of Mean 0.052 — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: Expansion Phase: Change From Baseline in Heart Rate at Week 20
Description: Heart rate was measured using electrocardiography. Least squares means are from a repeated measures model including treatment group, stratification factor, scheduled visit, interaction of treatment with scheduled visit and the baseline value as covariates.
Time Frame: Baseline and week 20
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 149 | 150 | 146
bpm | 0.57 (0.79) | -0.77 (0.79) | -2.40 (0.81)
Statistical Analysis 1: Comparison: Expansion Phase: Placebo vs Expansion Phase: Omecamtiv Mecarbil 25 mg; Test type: Other; p = 0.2177, Repeated Measures; Treatment difference = -1.34, 95% CI 2-sided [-3.47 to 0.79], Standard Error of Mean 1.09 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Expansion Phase: Placebo vs Expansion Phase: OM PK-based Titration; Test type: Other; p = 0.0070, Repeated Measures; Treatment difference = -2.97, 95% CI 2-sided [-5.12 to -0.81], Standard Error of Mean 1.09 — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: Expansion Phase: Change From Baseline in N-terminal Prohormone B-type Natriuretic Peptide (NT-proBNP) at Week 20
Description: Least squares means are from a repeated measures model including treatment group, stratification factor, scheduled visit, interaction of treatment with scheduled visit and the baseline value as covariates.
Time Frame: Baseline and week 20
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 149 | 150 | 146
pg/mL | 502 (257) | -319 (257) | -468 (262)
Statistical Analysis 1: Comparison: Expansion Phase: Placebo vs Expansion Phase: Omecamtiv Mecarbil 25 mg; Test type: Other; p = 0.0205, Repeated Measures; Treatment difference = -822, 95% CI 2-sided [-1516 to -127], Standard Error of Mean 353 — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Expansion Phase: Placebo vs Expansion Phase: OM PK-based Titration; Test type: Other; p = 0.0069, Repeated Measures; Treatment difference = -970, 95% CI 2-sided [-1672 to -268], Standard Error of Mean 357 — [estimate comment as in outcome 7, analysis 1]

13. Secondary Outcome: Dose Escalation Phase: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant, including worsening of a preexisting medical condition. The event does not necessarily have a causal relationship with study treatment. Laboratory value changes that required treatment or adjustment in current therapy were considered adverse events.
  Each adverse event was graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE), where Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = Severe AE, and Grade 4 = life-threatening AE.
  A serious adverse event is defined as an adverse event that met at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
Time Frame: From first dose of study drug to 4 weeks after last dose; treatment duration was 7 days in the dose escalation phase.
Population: Participants randomized in the dose-escalation phase who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Placebo | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Placebo | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2
Number analyzed (Participants) | 11 | 10 | 14 | 13 | 10 | 11 | 11 | 14
Participants
  Any treatment-emergent adverse event (TEAE) | 4 | 2 | 6 | 6 | 1 | 9 | 3 | 5
  TEAE Grade ≥ 2 | 0 | 1 | 1 | 1 | 1 | 5 | 1 | 1
  TEAE Grade ≥ 3 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
  TEAE Grade ≥ 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious adverse events | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
  TEAE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Fatal adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Expansion Phase: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a clinical trial participant, including worsening of a preexisting medical condition. The event does not necessarily have a causal relationship with study treatment. Laboratory value changes that required treatment or adjustment in current therapy were considered adverse events.
  Each adverse event was graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE), where Grade 1 = Mild AE, Grade 2 = Moderate AE, Grade 3 = Severe AE, and Grade 4 = life-threatening AE.
  A serious adverse event is defined as an adverse event that met at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * required in-patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
Time Frame: From first dose of study drug until 4 weeks after last dose; treatment duration was 20 weeks in the expansion phase.
Population: All participants randomized in the expansion phase who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Number analyzed (Participants) | 149 | 150 | 146
Participants
  Any treatment-emergent adverse event (TEAE) | 91 | 92 | 95
  TEAE Grade ≥ 2 | 62 | 60 | 61
  TEAE Grade ≥ 3 | 34 | 28 | 31
  TEAE Grade ≥ 4 | 5 | 8 | 11
  Serious adverse events | 30 | 36 | 32
  TEAEs leading to discontinuation of study drug | 12 | 8 | 12
  Fatal adverse events | 4 | 1 | 3

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 4 weeks after last dose; treatment duration was 7 days in the dose escalation phase and 20 weeks in the expansion phase.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Dose-escalation Cohort 1: Placebo: Participants received placebo tablets BID for 7 days.
Arm/Group | Dose-escalation Cohort 1: Placebo | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 | Dose-escalation Cohort 2: Placebo | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2 | Expansion Phase: Placebo | Expansion Phase: Omecamtiv Mecarbil 25 mg | Expansion Phase: OM PK-based Titration
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 1/14 | 0/13 | 0/10 | 2/11 | 0/11 | 1/14 | 30/149 | 36/150 | 32/146
Other Adverse Events (participants affected / at risk) | 4/11 | 2/10 | 5/14 | 6/13 | 1/10 | 8/11 | 3/11 | 4/14 | 48/149 | 51/150 | 48/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation Cohort 1: Placebo (N=11) | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 (N=10) | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 (N=14) | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 (N=13) | Dose-escalation Cohort 2: Placebo (N=10) | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 (N=11) | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 (N=11) | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2 (N=14) | Expansion Phase: Placebo (N=149) | Expansion Phase: Omecamtiv Mecarbil 25 mg (N=150) | Expansion Phase: OM PK-based Titration (N=146)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Cardiac asthma (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 5
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3
Cardio-respiratory distress (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation Cohort 1: Placebo (N=11) | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F1 (N=10) | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg M-F2 (N=14) | Dose-escalation Cohort 1: Omecamtiv Mecarbil 25 mg SCT-F2 (N=13) | Dose-escalation Cohort 2: Placebo (N=10) | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F1 (N=11) | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg M-F2 (N=11) | Dose-escalation Cohort 2: Omecamtiv Mecarbil 50 mg SCT-F2 (N=14) | Expansion Phase: Placebo (N=149) | Expansion Phase: Omecamtiv Mecarbil 25 mg (N=150) | Expansion Phase: OM PK-based Titration (N=146)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 2 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 3 | 4
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 5 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 8
Asthenia (General disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 14 | 9
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 8 | 5
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carotid bruit (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 9
Headache (Nervous system disorders) | 0 | 0 | 1 | 5 | 0 | 2 | 0 | 0 | 5 | 2 | 9
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 9 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 5
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.